CLINICAL TRIAL: NCT03153501
Title: How Should be Invasive Diagnostic Algorithm in Pleural Diseases
Brief Title: Efficiency and Safety of Pleural Biopsy Methods in the Diagnosis of Pleural Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eskisehir Osmangazi University (Other)
Responsible Party: Principal Investigator, Muzaffer Metintas, Medical Faculty, MD, Eskisehir Osmangazi University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PR-11-01-31-21
Record Dates: First submitted 2017-05-04; First posted 2017-05-15 (Actual); Last update posted 2017-05-15 (Actual); Status verified 2017-05

CONDITIONS: Diagnosis of Pleural Diseases; Medical Thoracoscopy

STUDY DESIGN:
Masking Description: Image guided biopsies Thoracoscopy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Diagnostic arm (Other): Patients with pleural diseases; malignant pleural diseases, tuberculous pleurisy, and other exudate required CT-guided Abrams needle biopsy, US-guided cutting needle biopsy, and medical thoracoscopy.
  Interventions: Diagnostic Test: CT-guided Abrams needle biopsy, US-guided cutting needle, medical thoracoscopy

INTERVENTIONS:
Diagnostic Test: CT-guided Abrams needle biopsy, US-guided cutting needle, medical thoracoscopy

SUMMARY:
Image-guided pleural biopsies, both ultrasound (US) or computed tomography (CT) guided, and medical thoracoscopy are important in the diagnosis of pleural disease. However, no consensus exists regarding which biopsy methods are appropriate for specific procedures.

In this prospective study, the investigators aimed to compare CT-scan guided pleural biopsy using an Abrams' needle (CT-ANPB) with US-assisted pleural biopsy using a cutting needle (US-CNPB)and medical thoracoscopy with respect to both diagnostic yield and safety.

DETAILED DESCRIPTION:
The primary end point of this study was the determination of the sensitivity and the complication rates of the invasive methods, Abrams needle pleural biopsy, tru-cut needle pleural biopsy, medical thoracoscopy with respect to the diagnosis of pleural disease.

ELIGIBILITY:
Inclusion Criteria:

* Patients with pleural diseases

Exclusion Criteria:

* Patients with other lung diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2011-02-08 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-04-30 (Actual)

PRIMARY OUTCOMES:
Diagnostic efficiencies of pleural biopsy methods; CT-guided Abrams needle, US-guided cutting needle and medical thoracoscopy in the diagnosis of pleural diseases: The sensitivity, specificity, negative predictive value and positive predictive value. | 5 years
  The sensitivity, specificity, negative predictive value and positive predictive value of computed tomography guided Abrams needle pleural biopsy, ultrasonography guided cutting needle biopsy and medical thoracoscopy techniques in the diagnosis of pleural diseases.
Safety of pleural biopsy methods; CT-guided Abrams needle, US-guided cutting needle and medical thoracoscopy in the diagnosis of pleural diseases: Rate of side effects. | 5 years
  Rate of side effects comparing to each other for computed tomography guided Abrams needle pleural biopsy, ultrasonography guided cutting needle biopsy and medical thoracoscopy techniques in the diagnosis of pleural diseases.

CONTACTS AND LOCATIONS:
Overall Officials: Muzaffer Metintas, MD, Principal Investigator — ESOGU Medical Faculty
Locations (2):
- Turkey (Türkiye) (2):
  - ESOGU Medical Faculty Department of Chest Diseases, Eskişehir, Meselik - Eskisehir
  - Eskisehir Osmangazi University Medical Faculty, Eskişehir

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim SJ, Choi SM, Lee J, Lee CH, Lee SM, Yim JJ, Yoo CG, Kim YW, Han SK, Park YS. Medical Thoracoscopy in Pleural Disease: Experience from a One-Center Study. Tuberc Respir Dis (Seoul). 2017 Apr;80(2):194-200. doi: 10.4046/trd.2017.80.2.194. Epub 2017 Mar 31. PMID 28416960